CLINICAL TRIAL: NCT01645059
Title: Observational, Cross-sectional, Multicenter Descriptive Study of the Patient Clinical Profile That Begins With Disseminated Her 2 + Breast Cancer or Develops a Metastasis After or During the Adjuvant Therapy (PRIMHER)
Brief Title: Multicenter Descriptive Study of the Patient Clinical Profile That Begins With Disseminated Her 2 + Breast Cancer or Develops a Metastasis After or During the Adjuvant Therapy
Acronym: PRIMHER
Status: Completed | Type: Observational
Sponsor: Asociación Cacereña para la Investigación y el Desarrollo en Oncología Médica (Network)
Responsible Party: Sponsor
Other Study IDs: ACI-CMM-2010-01
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-11

CONDITIONS: Disseminated HER2+ Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, cross-sectional study that the main objective is to describe the patient clinical profile that begins with disseminated Her 2+ Breast Cancer or develops a metastasis after or during the adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with 18 years or over
* Patients with disseminated breast cancer histologically or cytological confirmed, who begins with Her 2+ metastatic breast cancer or develops a metastasis after or during the adjuvant therapy
* Patients treated in first line treatment in metastatic disease.
* Patients who have positive Her 2 receptor test
* Patients who have given their written informed consent

Exclusion Criteria:

* Patients who are participating in other studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with disseminated HER2+ breast cancer in first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mª Helena López Ceballos, MD, Principal Investigator — Hospital San Pedro Alcántara; Santiago González Santiago, MD, Principal Investigator — Hospital San Pedro Alcántara
Locations (39):
- Spain (39):
  - Hospital de Denia, Denia, Alicante
  - Hospital General de Elda, Elda, Alicante
  - Hospital de Torrecárdenas, Almería, Almería
  - Hospital Infanta Cristina de Badajoz, Badajoz, Badajoz
  - Hospital don Benito, Don Benito, Badajoz
  - Hospital de Llerena, Llerena, Badajoz
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - ICO Badalona, Badalona, Barcelona
  - Clínica Corachan, Barcelona, Barcelona
  - Hospital General de l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital San Pedro Alcántara, Cáceres, Cáceres
  - Hospital Virgen del Puerto, Plasencia, Cáceres
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital de León, León, León
  - Hospital Universitario Arnau de Vilanova, Lleida, Lleida
  - Hospital Lucus Augusti, Lugo, Lugo
  - Hospital de Getafe, Getafe, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Morales Messeguer, Murcia, Murcia
  - Hospital Reina Sofía de Tudela, Tudela, Navarre
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital General de Segovia, Segovia, Segovia
  - Hospital Virgen de la Macarena, Seville, Sevilla
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital de Alcañiz, Alcañiz, Teruel
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Dr.Peset, Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid, Valladolid
  - Hospital Universitario Rio Hortega, Valladolid, Valladolid
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital de Zamora, Zamora, Zamora
  - Hospital de Txagorritxu, Vitoria-Gasteiz, Álava

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient included: 28th july 2011 Last Patient included: 27 th march 2013 Location: outpatient department
Period: Overall Study
Arm/Group | Disseminated Her 2+ Breast Cancer
Started | 129
Completed | 129
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Disseminated Her 2+ Breast Cancer
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 0
Region of Enrollment [Number; unit: participants]
  Spain | 129

OUTCOME MEASURES:

1. Primary Outcome: The Patient Clinical Profile (General Clinical Data and Breast Cancer Characteristics)
Description: General clinical data: age, weigh, height, Perfomance Status (ECOG Eastern Cooperative Oncology Group, runs from 0 to 5, with 0 denoting perfect health and 5 death), Breast cancer characteristics: familiar history of breast cancer, initial diagnostic (localized or disseminated), age at diagnostic, TNM (tumor node metástasis), tumor size, node involvement, primary tumor surgery, HER2 overexpression, histological Classification (grades I, II and III,determines the urgency and aggressiveness of treatment, as the higher grades do tend to correspond to poorer survival rates and prognosis), time from the primary breast cancer to distant relapse, description and localization of metastasis
Time Frame: 1 day (there is no follow-up, it is a cross-sectional study)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Disseminated Her 2+ Breast Cancer
Number analyzed (Participants) | 129
percentage of participants
  Perfomance Status (ECOG) 0 | 63.5 [54.4 to 71.8]
  Metastasic Breast Cancer | 48.8 [40.0 to 57.7]
  Ductal Carcinoma | 84.1 [76.3 to 89.8]
  Histological Grade III | 41.1 [32.6 to 50.1]
  Node involvement | 78.0 [69.3 to 84.9]
  Positive Estrogen Receptor | 57.5 [48.4 to 66.1]

2. Secondary Outcome: Adjuvant Treatment in Primary Breast Cancer: Chemotherapy (Treatment With TAC-Docetaxel, Adriamicine and Cyclophosphamide), Hormonal Therapy Anti-HER Biological Therapy
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Disseminated Her 2+ Breast Cancer
Number analyzed (Participants) | 66
percentage of participants
  Adjuvant treatment (Chemotherapy with TAC) | 22.0 [12 to 36.3]
  Adjuvant treatment (Hormonal therapy tamoxifen) | 41.7 [26.0 to 59.2]

3. Secondary Outcome: The Pattern of Treatment in Metastatic Breast Cancer: Chemotherapy, Hormonal Therapy Anti-HER Biological Therapy
Time Frame: one day (there is no follow-up, it si a cross-sectional study)
Measure: Number; unit: percentage of participants
Arm/Group | Disseminated HER 2 + Breast Cancer
Number analyzed (Participants) | 129
percentage of participants
  First line-Chemotherapy | 86.8
  Chemotherapy with Taxanes | 37.5
  Chemotherapy with Taxanes-Anthraciclines | 20.5
  Chemotherapy Vinorelbine | 17.0
  Hormonotherapy+ trastuzumab | 8.5
  Chemotherapy+ trastuzumab | 86.8

4. Secondary Outcome: Adjuvant Treatment and Age
Description: Adjuvant treatment and clinical profile (age)
  The patients analysed in this outcome are patients initially diagnosed with localized breast cáncer (N=66)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Trastuzumab Adjuvant Treatment | No Trastuzumab Adjuvant Treatment
Number analyzed (Participants) | 33 | 33
years | 55.3 (10.4) | 61.8 (13.4)

5. Secondary Outcome: Adjuvant Treatment-Physical Activity
Description: Adjuvant treatment and clinical profile (Physical activity)
  The patients analysed in this outcome are patients initially diagnosed with localized breast cáncer (N=66)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Number; unit: percentage of patients physical activity
Arm/Group | Trastuzumab Adjuvant Treatment | No Trastuzumab Adjuvant Treatment
Number analyzed (Participants) | 32 | 28
percentage of patients physical activity | 56.3 | 17.9

6. Secondary Outcome: Adjuvant Treatment-Node Affectation
Description: Adjuvant treatment and clinical profile (Node affectation)
  The patients analysed in this outcome are patients initially diagnosed with localized breast cáncer (N=66)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Number; unit: percentage of patients node affectation
Arm/Group | Trastuzumab Adjuvant Treatment | No Trastuzumab Adjuvant Treatment
Number analyzed (Participants) | 27 | 18
percentage of patients node affectation | 84.4 | 54.5

7. Secondary Outcome: Disseminated Breast Cancer Treatment-Age
Description: Analyse disseminated Breast Cancer treatment and clinical profile (age)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Taxanes First Line Treatment | No Taxanes First Line Treatment
Number analyzed (Participants) | 79 | 50
years | 56.1 (13.5) | 61.3 (14.1)

8. Secondary Outcome: Disseminated Breast Cancer Treatment-physical Activity
Description: Analyse disseminated Breast Cancer treatment and clinical profile (physical activity)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Number; unit: percentage of patients physical activity
Arm/Group | Taxanes First Line Treatment | No Taxanes First Line Treatment
Number analyzed (Participants) | 75 | 44
percentage of patients physical activity | 24 | 43.2

9. Secondary Outcome: Disseminated Breast Cancer Treatment-Smoking
Description: Analyse disseminated Breast Cancer treatment and clinical profile (Smoking)
Time Frame: one day (there is no follow-up, it is a cross-sectional study)
Measure: Number; unit: percentage of smoking participants
Arm/Group | Taxanes First Line Treatment | No Taxanes First Line Treatment
Number analyzed (Participants) | 76 | 47
percentage of smoking participants | 25 | 6.4

ADVERSE EVENTS:
Time Frame: 1 day
Description: Is a cross-sectional study
Arm/Group | Disseminated Her 2+ Breast Cancer
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 0/129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less